CLINICAL TRIAL: NCT01769313
Title: A Single Centre Study to Analyze Cataract Surgery Following Femtosecond Laser-Assisted and Manual Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1202
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Cataract
Keywords: Cataract; Laser-assisted; Femtosecond
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): In Group A the anterior capsulotomy and lens fragmentation will be performed by means of femtosecond laser surgery
  Interventions: Device: Laser-assisted cataract surgery
- Group B (Active Comparator): Group B acts as a control group where the capsulotomy as well as the lens fragmentation is performed manually.
  Interventions: Device: Manually performed cataract surgery

INTERVENTIONS:
Device: Laser-assisted cataract surgery — The anterior capsulotomy and lens fragmentation will be performed by means of femtosecond laser surgery
  Arms: Group A
Device: Manually performed cataract surgery — The anterior capsulotomy and lens fragmentation will be performed manually.
  Arms: Group B

SUMMARY:
This clinical study (non AMG/non MPG) is a contralateral, comparative, randomized, prospective, single-center, multi-surgeon, investigator masked study to investigate whether the femtolaser cataract surgery causes any significant differences in the resulting Intra Ocular Lens overlap (ΔROverlap) as compared to the conventional, manual continuous curvilinear capsulorhexis (CCC). The Intra Ocular Lens overlap (ΔROverlap) is defined as the difference between the Intra Ocular Lens center of mass to the capsulotomy aperture center of mass.

DETAILED DESCRIPTION:
A detailed pre-operative examination will ensure that every interested and willing patient fulfills the inclusion criteria of this study. For the proposed contralateral eye study between 30 and 35 patients will be enrolled whereas one eye will randomized undergo a manual cataract surgery and the other one a laser assisted cataract surgery. In total between 60 and 70 eyes will be included in the study. Pre-operative examinations are included to confirm to the clinical practice. Examinations on the day of surgery and any occurrence during the procedure are also listed. Post-operative examinations, which should document any occurrence, the outcome of and possible differences between the treatment techniques, are to be carried out after 1 day, 1 week, 1 month, 3 months and 6 months. After 6 month a final report including the study results will be produced.

The study is carried out in compliance with MEDDEV 2.7.1 Evaluation of Clinical Data: A Guide for Manufacturers and Notified Bodies, ICH E6 (R1) Good Clinical Practice (GCP), Declaration of Helsinki as well as the applicable local regulations such as notification requirements and current order of profession of the primary investigators.

ELIGIBILITY:
Inclusion Criteria:

* Clear corneal media
* Patients must be at least 18 years of age
* Patients must have read, understood and signed the Patient Information
* Patients are willing and able to return for follow-up examinations
* Topographic Astigmatism ≤ 1.5 dpt
* Patient will get a monofocal IOL (Envista) implanted

Exclusion Criteria:

* On a keratometric map of the cornea, the minimal and maximal K-values of the central 3mm zone must not differ by more than 5D (exclusion criterium for Group A only)
* The maximum K- value may not exceed 60D, the minimal value may not be smaller than 37D (exclusion criterium for Group A only)
* Corneal disease or pathology, such as corneal scaring or opacity, that precludes transmission of laser wavelength or that distorts laser light (exclusion criteria for Group A only)
* Subjects with a poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally
* Lens/zonular instability such as, but not restricted to, Marfan's Syndrome, Pseudoexfoliation Syndrome, etc.
* Manifest Glaucoma
* Patients presenting a clear lens (clear lens exchange)
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye
* Known sensitivity to planned concomitant medications
* Patients with disorders of the ocular muscle, such as nystagmus or strabismus
* Patients with keratoconus or keratectasia
* Patients with connective tissue weakness
* Patients who are blind on one eye
* Subjects who are immune compromised or carrying diagnosis of connective tissue disease, clinically significant atopic disease, insulin dependent diabetes mellitus, autoimmune diseases, ocular herpes zoster or simplex, endocrine diseases, lupus, rheumatoid arthritis, collagenosis and other acute or chronic illnesses that will increase the risk to the subject or confound the outcomes of this study.
* Abnormal examination results from slit lamp, fundus examination or IOL Master, age related changes are acceptable
* Abnormal examination results from Orbscan (exclusion criteria for Group A only; , age related changes are acceptable
* Patients who are pregnant or nursing
* Patients who do not give informed consent
* Patients with concentration disorders, epilepsy and other complicating diseases
* Patients regularly taking medicines that could influence the result of the treatment
* Patients who are participating in another ophthalmological clinical study
* Patients with an anterior chamber depth (ACD) < 1.5 mm or ACD > 4.8 mm as measured as from the corneal endothelium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
ΔROverlap is different between Group A and Group B | 6 Month postoeprative
  • The decentration, ΔROverlap, between implanted IOL and capsulotomy aperture is different in Group A as compared to Group B. p<0.05 will be considered statistically significant.
  The study end point will be determined for all follow-up examination periods; the purpose criterion should be achieved by the 6 month examination at the latest.
  Goal:To evaluate a significant difference (p<0.05) of ΔROverlap between Group A and Group B

SECONDARY OUTCOMES:
ΔELP is different between Group A and Group B | 6 months postoperative
  • The difference, Δ Flare, between preoperative and postoperative is different for Group A as compared to group B. p<0.05 will be considered statistically significant.
  The study end point will be determined 1-Day and 1-Week follow-up examination periods; the purpose criterion should be achieved by the 1-Week follow-up examination at the latest.
  Goal:
  To evaluate a significant difference (p<0.05) of Δ Flare between Group A and Group B
ΔFlare is different between Group A and Group B | 6 months postoperative
  • The difference, Δ Flare, between preoperative and postoperative is different for Group A as compared to group B. p<0.05 will be considered statistically significant.
  The study end point will be determined 1-Day and 1-Week follow-up examination periods; the purpose criterion should be achieved by the 1-Week follow-up examination at the latest.
  Goal:
  To evaluate a significant difference (p<0.05) of Δ Flare between Group A and Group B
SEQ Prediction Error is different between Group A and Group B | 6 months postoperatvie
  • The difference, SEQ Prediction Error, between target refraction SEQ and actual SEQ is different in Group A as compared to Group B. p<0.05 will be considered statistically significant.
  The study end point will be determined for all follow-up examination periods, the purpose criterion should be achieved by the 6 month examination at the latest.
  Goal:
  To evaluate a significant difference (p<0.05) of the SEQ Prediction Error between Group A and Group B

CONTACTS AND LOCATIONS:
Overall Officials: Gerd U Auffarth, Prof. Dr., Principal Investigator — Universitäts-Augenklinik Heidelberg
Locations (1):
- Universitäts-Augenklinik Heidelberg, Heidelberg, Germany